CLINICAL TRIAL: NCT03121729
Title: Enhanced Recovery After Surgery Program for Gastric Cancer: a Multi-center Study
Acronym: ERASG1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jian ZHAO, Vice director of Research Institute of General Surgery, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BE2015687
Record Dates: First submitted 2017-04-13; First posted 2017-04-20 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Gastric Cancer
Keywords: enhanced recovery after surgery; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Intervention Model Description: Patients will receive enhanced recovery after surgery programs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- enhanced recovery after surgery (Experimental): enhanced recovery after surgery includes:
  1. Multimodal analgesia
  2. Early oral intake A: Drink water after anesthetic awareness. B: Recover semi-liquid diet
  3. Management of nasogastric tube and catheter A: Not indwell nasogastric tube conventionally B: Remove catheter early
  4. Early activity
  5. Perioperative controlled infusion A: Load carbohydrate preoperatively B: No preoperative bowel preparation C: Fast six hours before surgery, no drink two hours before surgery D: Intraoperative liquid management: 3-6ml/kg/h, determined by anesthetists E: Stop intravenous infusion upon 2000-2500ml water and semiliquid diet being taken
  Interventions: Procedure: enhanced recovery after surgery

INTERVENTIONS:
Procedure: enhanced recovery after surgery — Undergo an enhanced recovery after surgery program

SUMMARY:
This study is aimed to evaluate the safety of applying enhanced recovery after surgery for gastric cancer.

DETAILED DESCRIPTION:
In China, gastric cancer results in the second highest morbidity and mortality rates among all malignancies. It is very important for treatment of gastric cancer to enhance the quality of treatment, increase patients' survival rate and improve the life quality. Now, "Gastric Cancer, Version 3.2016, NCCN Clinical Practice Guidelines in Oncology" and "Japanese gastric cancer treatment guidelines 2014 (ver. 4)" recommended surgical resection for gastric cancer. As a result, increasing the quality of surgery and improving the perioperative measures have a great influence on patients received a gastrectomy. Before, patients discharged on 7-10 days after gastrectomy and recovered 4-8 weeks after surgery. So, it is significant for patients to recover from surgical trauma in order to receive other anti-cancer therapies after gastrectomy. Investigators spent over ten years studying enhanced recovery after surgery programs for gastric cancer and have got some successful experience. Investigators found enhanced recovery after surgery can accelerate patients' recovery without increasing complications.

This study is the first multi-center study of enhanced recovery after surgery for gastric cancer all over the world. During this period, the study is aimed to evaluate the safety of applying enhanced recovery after surgery for gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Requirements of informed consent and assent of participant, parent or legal guardian as applicable
2. Patients with gastric cancer scheduled for radical gastrectomy and between the age of 18 and 75 years old without considering sex
3. ASA physical status I-III
4. Participants can follow the drug doses and visit plan

Exclusion Criteria:

1. Patients certified by a doctor that doesn't fit to participate in this study.
2. Patients with ischemic heart disease, cerebrovascular disease and peripheral vascular disease, or their cardiac function > II (NYHA) patients, patients received CABG recently, and patients with severe hypertension (systolic pressure≥180mmHg or diastolic pressure≥110mmHg).
3. Patients with gastric cancer with distant metastasis.
4. Patients with severe infection, respiratory dysfunction, coagulation disorders, severe liver and renal dysfunction (Child - Pugh≥ 10; creatinine clearance < 25 ml/min).
5. Patients allergic to common drugs, such as opioids, non-steroidal drugs, cephalosporins, etc.
6. Patients with operations of gastrointestinal cancer and complicated abdominal operations.
7. Patients complicated by gastric cancer with complications such as hemorrhage, perforation, obstruction.
8. Patients with dyscrasia and severe malnutrition (albumin≤30g/L, weight loss in half a year>10%, SGA classification C, BMI<18, Hb<70g/L).
9. Patients with metabolic complications caused by diabetes.
10. Patients can't finish enhanced recovery after surgery programs and have contraindications of enhanced recovery after surgery.
11. Pregnancy and lactation women, or have a pregnancy plan within a month after the test of the subjects (also including male participants).
12. Patients participated other subjects 3 months before this subject.
13. Sponsors or researchers directly involved in the testing or their family members.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-06-21 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
occurrence rate of severe complications | 1 month
  including death, anastomotic fistula, intra-abdominal hemorrhage, hemorrhage of digestive tract and complications need a reoperation

SECONDARY OUTCOMES:
Occurrence rate of ordinary complications | 1 month
  Except severe complications, Clavien-Dindo classification ≥Ⅱ complications need not reoperation
Readmission rate within 30 days after discharge | 1 month
  Readmission rate within 30 days after discharge
Ideal postoperative length of hospital stay | 1 month
  reach discharge criteria
Actual postoperative length of hospital stay | 1 month
  Actual postoperative length of hospital stay
Operative time | 1 day
  Data of operation
Blood loss | 1 day
  Data of operation
Intraoperative infusion | 1 day
  Data of operation
TNM classification | 1 week
  Data of tumor
Number of dissected lymph node | 1 week
  Data of tumor
Time to first flatus | 2 week
  Bowel function recovery
Time to first defecation | 2 week
  Bowel function recovery
Time to first semi-liquid diet | 2 week
  Bowel function recovery
Time to first off-bed activity | 1 week
  Postoperative activity
Time of off-bed activity per day | 1 week
  Postoperative activity
Distance of off-bed activity per day | 1 week
  Postoperative activity
Postoperative pain | 1 week
  VAS classification
Hospital cost | 1 month
  Hospital cost
Management of catheters | 1 month
  including nasogastric tube, catheter, intraperitoneal drain, infusion tube
Preoperative length of hospital stay | 1 month
  Preoperative length of hospital stay
CD3+ | 1 week
  Immune indicators
CD4+ | 1 week
  Immune indicators
CD4+/CD8+ | 1 week
  Immune indicators
IL-6 | 1 week
  Inflammatory indicators
CRP | 1 week
  Inflammatory indicators
Albumin | 1 week
  Nutritional indicators
Prealbumin | 1 week
  Nutritional indicators
Transferrin | 1 week
  Nutritional indicators
Hb | 1 week
  Nutritional indicators
WBC | 1 week
  Nutritional indicators
PLT | 1 week
  Nutritional indicators
HCT | 1 week
  Nutritional indicators
Blood glucose | 1 week
  Nutritional indicators
Procalcitonin | 1 week
  Infectious indicator

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Wei JIANG, Ph.D., Principal Investigator — Jinling Hospital, Medical School of Nanjing University; Jian ZHAO, Ph.D., Study Director — Jinling Hospital, Medical School of Nanjing University; Gang WANG, Ph.D., Study Director — Jinling Hospital, Medical School of Nanjing University; Jiang LIU, M.D., Study Director — Jinling Hospital, Medical School of Nanjing University
Locations (23):
- China (23):
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Changzhou Second People's Hospital Affiliated to Nanjing Medical University, Changzhou, Jiangsu
  - The First People's Hospital of Lianyungang City, Lianyungang, Jiangsu
  - The Second People's Hospital of Lianyungang City, Lianyungang, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Jinling Hospital, Medical School of Nanjing University, Nanjing, Jiangsu
  - Zhongda Hospital, Southeast University, Nanjing, Jiangsu
  - the Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Suqian People's Hospital, Nanjing Drum Tower Hospital, Suqian, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First People's Hospital of Taicang, Suzhou, Jiangsu
  - Zhangjiagang First People's Hospital, Suzhou, Jiangsu
  - the Taizhou People's Hospital, Taizhou, Jiangsu
  - The 101 Hospital of the Chinese People's Liberation Army, Wuxi, Jiangsu
  - Affiliated Hospital of Jiangnan University, The Forth People's Hospital of Wuxi City, Wuxi, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Affiliated People's Hospital of Jiangsu University, Zhenjiang, Jiangsu

IPD SHARING:
Plan to Share IPD: No